CLINICAL TRIAL: NCT03515109
Title: Prospective Randomized Trial of Altis Minisling With the TVTO Transobturator Tape Procedure for the Management of Genuine Stress Urinaty Incontinence in Women
Brief Title: Prospective Study of Altis System With the TVTO Procedure for the Management of Stress Urinary Incontinence in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieio Hospital (Other)
Responsible Party: Principal Investigator, PANAGIOTIS BAKAS MD, Associate Professor Obstetrics and Gynecology, Aretaieio Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2018-03-23; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Genuine Stress Incontinence
Keywords: stress incontinence; female; altis; transobturator tape; minisling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: prospective randomised
Who Masked: Participant, Investigator
Masking Description: they will not be aware of the procedure they are going to perform or have.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- group A (Active Comparator): Altis tape surgical placement
  Interventions: Procedure: Altis tape
- group B (Placebo Comparator): TVT transobturator tape placement
  Interventions: Procedure: TVTO

INTERVENTIONS:
Procedure: Altis tape — placement of Altis tape through transobturator foramen bilaterally under epidural anesthesia
  Arms: group A
Procedure: TVTO — placement of TVTO tape through transobturator foarmen bilaterally under epidural anesthesia
  Arms: group B

SUMMARY:
Prospective randomized comparison of minisling (altis) with the TVTO procedure for the management of women with genuine stress urinary incontinence.

DETAILED DESCRIPTION:
Prospective randomized study double blinded. Two group of patients consisting group A of 40 patients being operated with altis minisling and group B with 40 patients operated with TVTO procedure. All patients will be operated with epidural anesthesia.

The patients participating in the study will meet the following requirements. a. Having genuine stress urinary incontinence proven by urodynamics, b. be willing to be operated and participate in the study. Exclusion criteria wil be the following: a.History of previous irradiation in the lower genital tract, b. BMI more than 30kg/m2, c.previous anti-incontinence surgery, previous vaginal surgery, e. having MUCP< 20 cm H2O or Valsava leak point pressure less than than 60 cm H2O.

Patients will be allocated in each operation by an automatic system using a computer software.

Primary outcome measure will be the objective cure rate at 6 months as it is assessed with cough stress test during urodynamics. Secondary outcome measures will be the subjective cure rate, improvement and failure rate, the incidence of complications such as obstruction, voiding difficulties, hemorrhage etc. Patients will be asked to complete preoperatively and postoperatively the ICIQ-FLUTS, patient satisfaction questionnaire and the female sexual function index.postoperatively the patients will complete the PGI-I questionnaire.

ELIGIBILITY:
Inclusin Criteria:

* Having genuine stress urinary incontinence proven by urodynamics
* be willing to be operated and participate in the study.

Exclusion Criteria:

* History of previous irradiation in the lower genital tract
* BMI more than 30kg/m2
* previous anti-incontinence surgery, previous vaginal surgery
* having MUCP< 30 cm H2O or Valsava leak point pressure less than than 60 cm H2O
* Mixed urinary incontinence.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2018-11-25 (Estimated)

PRIMARY OUTCOMES:
the objective urinary continence rate at 12 months | 1 year
  Primary outcome measure will be the objective urinary continence rate at 12 months as it is assessed with cough stress test during urodynamics.

SECONDARY OUTCOMES:
Subjective urinary continence rate at 12 months follow up | 1year
  Secondary outcome measure will be the subjective continence rate as it is assessed with the use of the PGI-I questionnaire.
Preoperative and postoperative assessment of sexual function | 1 year
  Patients will be asked to complete preoperatively and postoperatively the female sexual function index. Minimum score 2.0 and maximum score 36.0. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: PANAGIOTIS VAKAS, Principal Investigator — aretaieio university hospital
Locations (1):
- Aretaieio University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839